CLINICAL TRIAL: NCT05201404
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Namodenoson in the Treatment of Advanced Hepatocellular Carcinoma in Patients With Child-Pugh Class B7 Cirrhosis
Brief Title: Namodenoson in the Treatment of Advanced Hepatocellular Carcinoma in Patients With Child-Pugh Class B7 Cirrhosis
Acronym: LIVERATION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF102-301HCC
Record Dates: First submitted 2021-12-21; First posted 2022-01-21 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
Keywords: Hepatocellular carcinoma; HCC; Liver cancer; Child-Pugh Class B7 cirrhosis; CPB7
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Liver Neoplasms | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Intervention Model Description: Parallel group, double-blinded, randomization in a 1:1 ratio to active versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Namodenoson (CF102) (Experimental): Namodenoson 25 mg orally BID, until disease progression or unacceptable adverse events
  Interventions: Drug: Namodenoson
- Placebo (Placebo Comparator): Matching placebo orally BID, until disease progression or unacceptable adverse events
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Namodenoson — Adenosine A3 Receptor (A3AR) agonist
  Other Names: CF102
  Arms: Namodenoson (CF102)
Drug: Placebo — Control arm
  Other Names: Inactive control
  Arms: Placebo

SUMMARY:
This is a clinical trial in patients with advanced hepatocellular carcinoma (HCC) and Child-Pugh Class B7 (CPB7) cirrhosis whose disease has progressed on at least 1st-line therapy. The trial will evaluate the efficacy and safety of namodenoson as compared to placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial in patients with advanced HCC and CPB7 cirrhosis whose disease has progressed on at least 1st-line therapy. The trial will evaluate the efficacy and safety of namodenoson as compared to placebo. Patients will be randomly assigned in a 2:1 ratio to treatment with oral doses of either namodenoson 25 mg or matching placebo administered twice daily for consecutive 28-day cycles. Patients will be evaluated regularly for safety. Tumor imaging will be performed every two cycles. Treatment will continue until the patient experiences PD or unacceptable drug-related intolerability. Patients will return for a follow-up visit 28 days after completion of the last dose of study drug, and survival data will be obtained for all randomized patients who consent to long-term follow-up. Patients who discontinue dosing and consent to follow-up will be followed indefinitely for survival status.

Once the requisite number of events has been observed and the blind is broken for analysis of the trial results, any surviving patients who remain on blinded drug will be offered the opportunity to continue dosing with OL namodenoson 25 mg twice daily indefinitely.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Diagnosis of HCC:

   * For patients without cirrhosis at the time of diagnosis, histologic confirmation is required (archival tissue is acceptable).
   * For patients with underlying cirrhosis at the time of diagnosis, diagnosis of HCC established according to the American Association for the Study of Liver Diseases Practice Guideline algorithm (Marrero 2018).
3. HCC is advanced (i.e., treatment-refractory or metastatic) and no standard therapies are expected to be curative.
4. HCC has progressed on at least 1, but no more than 2, prior systemic treatment regimens; prior locoregional therapy is allowed.
5. Barcelona Clinic Liver Cancer (BCLC) Stage B or C (Llovet 1999).
6. Prior HCC treatment was discontinued for at least 2 weeks prior to the Baseline Visit.
7. Measurable disease by RECIST v1.1 (Eisenhauer 2009).
8. ECOG PS of ≤ 1.
9. Cirrhosis classified as CPB7; if ascites is used as a scoring criterion, it must be classified as Grade ≥2 by the Clinical Practice Guidelines of the European Association for the Study of the Liver (EASL 2010).
10. The following laboratory values must be documented within ten days prior to the first dose of study drug:

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
    * Platelet count at least 75 × 10^9/L
    * Creatinine clearance at least 50 mg/dL (estimated glomerular filtration rate by the Cockcroft-Gault or the Modification of Diet in Renal Disease methods)
    * AST and ALT ≤ 5 × the upper limit of normal (ULN)
    * Total bilirubin ≤ 3.0 mg/dL
    * Serum albumin ≥ 2.8 g/dL.
11. Life expectancy of ≥ 6 weeks.
12. For women of childbearing potential, negative serum pregnancy test result.
13. Provide written informed consent to participate.
14. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other trial-related procedures.

Exclusion Criteria:

1. Receipt of >2 prior systemic drug therapies for HCC.
2. Receipt of systemic cancer therapy, immunomodulatory drug therapy, immunosuppressive therapy, or corticosteroids > 20 mg/day prednisone or equivalent within 14 days prior to the Baseline Visit or concurrently during the trial.
3. Locoregional treatment within 4 weeks prior to the Baseline Visit.
4. Major surgery or radiation therapy within 4 weeks prior to the Baseline Visit.
5. Use of any investigational agent within 4 weeks prior to the Baseline Visit.
6. Concomitant use of P-glycoprotein (P-gp)/breast cancer resistance protein (BCRP) inhibitors and/or substrates with a narrow therapeutic index unless the medication can be taken at least 3 hours before or after taking the investigational product (see Section 12.2).
7. Child-Pugh Class A, B8/9, or C cirrhosis.
8. Hepatic encephalopathy.
9. Occurrence of esophageal or other gastrointestinal hemorrhage requiring transfusion within 4 weeks prior to the Baseline Visit.
10. Uncontrolled or clinically unstable thyroid disease, per judgment of the Principal Investigator.
11. Active bacterial, viral, or fungal infection requiring systemic therapy or operative or radiological intervention.
12. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
13. Liver transplant.
14. Active malignancy other than HCC.
15. Uncontrolled arterial hypertension or congestive heart failure (New York Heart Association Classification 3 or 4).
16. Angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
17. History of, or ongoing, cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 470 msec (patients with bundle branch block will not be excluded for QTc reasons).
18. Pregnant or lactating female.
19. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Investigator, are effective and adequate for the patient's circumstances while on study drug.
20. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug and for 3 months afterward.
21. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with trial participation or study drug administration; may interfere with the informed consent process and/or with compliance with the requirements of the trial; or may interfere with the interpretation of trial results and, in the Investigator's opinion, would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the time of randomization until the date of death from any cause, assessed up to 60 months
  Median duration of survival

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the time of randomization until the date of disease progression or death from any cause, assessed up to 60 months
  Median time to disease progression using RECIST and modified RECIST criteria
Objective Response Rate (ORR) | Through study completion, with a median of 9 months
  Proportion of patients who experience Objective Response (OR) using RECIST and modified RECIST criteria
Incidence and nature of treatment-emergent adverse events | Through study completion, with a median of 9 months
  Incidence and nature of treatment-emergent adverse events as assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v5)
Pharmacokinetics (PK) of namodenoson in this population | 29 days
  Plasma concentration of namodenoson

OTHER OUTCOMES:
Duration Of Response (DOR) | Through study completion, with median of 9 months
  Time from first response (CR or PR) to progression or death, whichever occurs first
Disease Control Rate (DCR) | Through study completion, with median of 9 months
  Proportion of patients who experience OR as well as those who experience Stable Disease (SD) for at least four treatment cycles, ie, four months
Quality of Life (QOL) using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) | Through study completion, with a median of 9 months
  Assess QOL in this population using the EORTC QLQ-C30, a 30-item questionnaire. Each question is measured in a range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life (QOL), using the hepatocellular carcinoma- (HCC-) specific module of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Hepatocellular Carcinoma 18-question Module (EORTC QLQ-HCC18) | Through study completion, with a median of 9 months
  Assess QOL in this population using the HCC-specific module of the EORTC QLQ-HCC18, an 18-item questionnaire. Each question is measured in a range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (32):
- Site 881, Dallas, Texas, United States
- Bosnia and Herzegovina (3):
  - 841 University Clinical Centre of Republic of Srpska, Banja Luka
  - 843 University Clinical Hospital Mostar, Mostar
  - 842 University Clinical Centre Sarajevo, Sarajevo
- Bulgaria (4):
  - 831 Dept of Medical Oncology, Complex Oncology Ctr - Burgas EOOD, Burgas
  - 835 First Department of Medical Oncology, Gastroenterology and Pulmology, Complex Oncology Center - Plovdiv EOOD, Plovdiv, Plovdiv
  - Medical Center Leo Clinic EOOD Plovdiv, Plovdiv
  - 834 Medical Oncology Dept, Univ Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski" EAD, Sofia, Sofia
- 518 Rabin Medical Center Beilinson Hospital, Petah Tikva, Israel
- 872 IMSP Institute of Oncology, Chisinau, Moldova
- Poland (6):
  - Site 858, Koszalin
  - Site 852, Krakow
  - Site 857, Mysłowice
  - Site 859, Przemyśl
  - Site 855, Warsaw
  - Site 850, Wroclaw
- Romania (10):
  - 802 Institutul Regional de Gastroenterologie si Hepatologie, Cluj-Napoca
  - 807 IOCN, Medical Oncology, Cluj-Napoca
  - 809 Spitalul Clinic Judetean de Urgenta Constanta Oncology Dept, Constanța
  - 801 Oncology Center "Sf. Nectarie" Medical Oncology, Craiova
  - 803 Oncolab SRL, Craiova
  - 805 Euroclinic lasi, Iași
  - 810 IRO Iasi-Clinica Oncologie Medicala, Iași
  - 808 Spitalul Clinic Pelican Oradea Oncology Department, Oradea
  - 804 Oncomed - Medical Oncology, Timișoara
  - 806 Oncocenter Oncologie Clinica SRL, Timișoara
- Serbia (4):
  - 821 Clinic for Gastroenterology and Hepatology, Military Medical Academy, Belgrade
  - 822 Oncology Institute of Vojvodina, Kamenitz
  - 823 Oncology Department, Health Center Kladovo, Kladovo
  - 824 Univ Clin Centre Kragujevac, Dept of Oncology, Kragujevac
- Slovakia (2):
  - Site 867, Banská Bystrica
  - Site 865, Košice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bar-Yehuda S, Stemmer SM, Madi L, Castel D, Ochaion A, Cohen S, Barer F, Zabutti A, Perez-Liz G, Del Valle L, Fishman P. The A3 adenosine receptor agonist CF102 induces apoptosis of hepatocellular carcinoma via de-regulation of the Wnt and NF-kappaB signal transduction pathways. Int J Oncol. 2008 Aug;33(2):287-95. PMID 18636149
- [Background] Cohen S, Stemmer SM, Zozulya G, Ochaion A, Patoka R, Barer F, Bar-Yehuda S, Rath-Wolfson L, Jacobson KA, Fishman P. CF102 an A3 adenosine receptor agonist mediates anti-tumor and anti-inflammatory effects in the liver. J Cell Physiol. 2011 Sep;226(9):2438-47. doi: 10.1002/jcp.22593. PMID 21660967
- [Background] Stemmer SM, Benjaminov O, Medalia G, Ciuraru NB, Silverman MH, Bar-Yehuda S, Fishman S, Harpaz Z, Farbstein M, Cohen S, Patoka R, Singer B, Kerns WD, Fishman P. CF102 for the treatment of hepatocellular carcinoma: a phase I/II, open-label, dose-escalation study. Oncologist. 2013;18(1):25-6. doi: 10.1634/theoncologist.2012-0211. Epub 2013 Jan 8. PMID 23299770
- [Background] Stemmer SM, Manojlovic NS, Marinca MV, Petrov P, Cherciu N, Ganea D, Ciuleanu TE, Pusca IA, Beg MS, Purcell WT, Croitoru AE, Ilieva RN, Natosevic S, Nita AL, Kalev DN, Harpaz Z, Farbstein M, Silverman MH, Bristol D, Itzhak I, Fishman P. Namodenoson in Advanced Hepatocellular Carcinoma and Child-Pugh B Cirrhosis: Randomized Placebo-Controlled Clinical Trial. Cancers (Basel). 2021 Jan 7;13(2):187. doi: 10.3390/cancers13020187. PMID 33430312
- See also: Sponsor website — https://www.canfite.com/